CLINICAL TRIAL: NCT05767866
Title: Safety and Preliminary Efficacy of YK-029A, a Novel EGFR TKI, in Patients With Advanced NSCLC Harboring ex20ins, T790M or Rare Mutations
Brief Title: Assessing an Oral EGFR Inhibitor,YK-209A in Patients Who Have Advanced Non-small Cell Lung Cancer With EGFR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Puhe Pharmaceutical Technology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNYK-01
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Treatment; Treatment Side Effects
Keywords: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part 1: Dose Escalation Component (Experimental): In dose-escalation phase, previously treated patients with EGFR T790M mutation were enrolled. YK-029A was given at doses of 50, 100, 150, 200 to 250 mg/day (3+3 design).
  Interventions: Drug: YK-029A
- Part 2: Expansion Cohort 1 (Experimental): In dose-escalation phase, previously treated patients with EGFR T790M mutation were enrolled. YK-029A was given at doses of 50mg/day and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A
- Part 2: Expansion Cohort 2 (Experimental): In dose-escalation phase, previously treated patients with EGFR T790M mutation were enrolled. YK-029A was given at doses of 100mg/day and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A
- Part 2: Expansion Cohort 3 (Experimental): In dose-escalation phase, previously treated patients with EGFR T790M mutation were enrolled. YK-029A was given at doses of 150mg/day and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A
- Part 3: ExTension Cohort 4 (Experimental): In dose-extension phase, previously treated patients with EGFR exon 20ins mutation were enrolled. YK-029A was given at doses of 150mg/day and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A
- Part 3: ExTension Cohort 5 (Experimental): In dose-extension phase, previously treated patients with EGFR exon 20ins mutation were enrolled. YK-029A was given at doses of 200mg/day and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A
- Part 3: ExTension Cohort 6 (Experimental): In dose-extension phase, previously untreated patients with EGFR exon 20ins mutation were enrolled. YK-029A was given at doses of 200mg/day and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A
- Part 3: ExTension Cohort 7 (Experimental): In dose-extension phase, previously treated patients with EGFR rare mutation （G719X、L861Q、S768I etal.)were enrolled. YK-029A was given at doses of 150mg/day and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A
- Part 3: ExTension Cohort 8 (Experimental): In dose-extension phase, previously treated patients with EGFR rare mutation （G719X、L861Q、S768I etal.)were enrolled. YK-029A was given at doses of 200mg/day and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A
- Part 3: ExTension Cohort 9 (Experimental): In dose-extension phase, previously untreated patients with EGFR exon 20ins mutation were enrolled. YK-029A was given at doses of 150mgBID and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: YK-029A

INTERVENTIONS:
Drug: YK-029A — Daily dose of YK-029A

SUMMARY:
This study aimed to evaluate the safety and preliminary efficacy of YK-029A, a novel third-generation epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor, in treated or untreated patients with advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This phase 1/2 study will evaluate the safety, pharmacokinetics, and anti-tumor activity of oral EGFR Inhibitor YK-209A in participants with NSCLC and anti-tumor activity of YK-029A in participants with solid tumors other than NSCLC harboring ex20ins, T790M or rare mutations. The trial will be conducted in three parts: a dose escalation (Part 1), expansion phase (Part 2), followed by an extension phase (Part 3).

The objectives of the dose escalation phase (Part 1), is to determine the safety profile of orally administered YK-029A, including the MTD, DLTs, RP2D, pharmacokinetic profile. The primary goal of the expansion component of the trial is to evaluate the anti-tumor activity of YK-029A in nine histologically and molecularly defined cohorts at the RP2D (determined based on dose escalation phase of the trial).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria all cohorts: dose escalation, dose expansion, and dose extension:

1. Have histologically or cytologically confirmed locally advanced or metastatic NSCLC disease (Stage IIIB or IV) .
2. Male or femal adult，be able to provide a signed and dated, written informed consent.
3. Must have measurable disease by response evaluation criteria in solid tumors (RECIST) v1.1.
4. Minimum life expectancy of 3 months or more.
5. Adequate organ function at baseline.
6. Normal QT interval on screening electrocardiogram (ECG), defined as QT interval corrected (Fridericia) (QTcF) of less than or equal to (≤ ) 450 millisecond (ms) in males or ≤ 470 ms in females.

Part 1: Dose Escalation Cohort Specific Inclusion Criteria:

1. Refractory to standard available therapies.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
3. aged 18-65 years old.
4. previously treated NSCLC patients with EGFR T790M.

Part 2: Expansion Cohort 1、2、3 Specific Inclusion Criteria:

1. previously treated NSCLC patients with EGFR T790M.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
3. aged 18-75 years old.

Part 2: Expansion Cohort 4、5 Specific Inclusion Criteria:

1. previously treated NSCLC patients with EGFR exton 20ins.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
3. aged 18-75 years old.

Part 3: Expansion Cohort 6 Specific Inclusion Criteria:

1. previously untreated NSCLC patients with EGFR exton 20ins.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
3. aged 18-75 years old.

Part 3: Expansion Cohort 7、8 Specific Inclusion Criteria:

1. previously treated NSCLC patients with EGFR rare mutation(（G719X、L861Q、S768I).
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
3. aged 18-75 years old.

Part 3: Expansion Cohort9 Specific Inclusion Criteria:

1. previously treated NSCLC patients with EGFR exton 20ins.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
3. aged 18-75 years old.

Exclusion Criteria:

1. Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days before screening.
2. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose or with a wide field of radiation which must be completed within 4 weeks before screening.
3. NSCLC patients with EGFR T790M mutation previously treated with third-generation EGFR-TKIs (such as AZD9291, CO-1686, HM61713, EGF816, PF-06747775, vometinib, BPI-15086, Ivirtinib maleate, etc.) and their apis or the same drugs in other clinical trials Drug treatment.
4. Patients with NSCLC with EGFR ex20ins mutation had previously received EGFR ex20ins inhibitors and/or EGFR-cMET double antibodies (including but not limited to TAK-788, bociotinib, JNJ-61186372, DZD9008, vometinib, PLB1004, and AZD9291 in excess of the clinically approved dose (cohort 9 prohibited AZD9291 at any dose) and Drug substance or other similar drug treatment in the clinical trial stage.
5. NSCLC patients with rare EGFR mutations have previously been treated with third-generation EGFR-Tkis (such as AZD9291, etc.) and their apis or other similar drugs in clinical trials.
6. Received a moderate or strong CYP4503A inhibitor or moderate or strong CYP3A inducer within 10 days prior to first dose of YK-029A.
7. Have significant, uncontrolled, or active cardiovascular disease.
8. Have a known history of uncontrolled hypertension. Participants with hypertension should be under treatment on study entry to control blood pressure.
9. Have prolonged QTcF interval, or being treated with medications known to be associated with the development of torsades de pointes.
10. Have an ongoing or active infection, including but not limited to, the requirement for intravenous (IV) antibiotics, or a known history of human immunodeficiency virus, hepatitis B virus (HBV), or hepatitis C virus (HCV). Testing is not required in the absence of history.
11. Currently have or have a history of interstitial lung disease, radiation pneumonitis that required steroid treatment, or drug-related pneumonitis.
12. Female participants who are lactating and breastfeeding or have a positive urine or serum pregnancy test during the screening period.

    Note: Female participants who are lactating will be eligible if they discontinue breastfeeding.
13. Have gastrointestinal illness or disorder that could affect oral absorption of YK-029A.
14. Have any condition or illness that, in the opinion of the investigator, might compromise participant safety or interfere with the evaluation of the safety of the drug.
15. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-75 Years and older (Adult, Older Adult)
Enrollment: 160 (Estimated)
Dates: Start 2018-03-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants that Experience Adverse Events (AEs) and Serious Adverse Events (SAEs) . | Cycle 1 (Cycle length is equal to [=] 28 days)
  To investigate the safety and tolerability of YK-029A when given orally to patients with advanced NSCLC with EGFR T790M.
Part 1: Number of Participants with Clinically Significant Abnormal Laboratory Values. | Cycle 1 (Cycle length is equal to [=] 28 days)
  To investigate the safety and tolerability of YK-029A when given orally to patients with advanced NSCLC with EGFR T790M.
Part 1: Number of Participants with First Cycle Dose-Limiting Toxicities (DLTs). | Cycle 1 (Cycle length is equal to [=] 28 days)
  To establish Maximum Tolerated Dose (MTD) (if possible) and Recommended Phase 2 Dose (PR2D) of YK-029A when given orally in patients with advanced NSCLC with EGFR T790M mutations.
Part 1: DLTs of Orally Administered YK-029A. | Cycle 1 (Cycle length is equal to [=] 28 days)
  Toxicity will be Evaluated According to the NCI CTCAE, Version 5.00. DLT will be defined as any of the events specified in the protocol that are considered by the investigator to be at least possibly related to therapy with study medications.
Part 1: Number of Participants with First Cycle Dose-Limiting Toxicities (DLTs). | Cycle 1 (Cycle length is equal to [=] 28 days)
  Toxicity will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.00. DLT will be defined as any of the events specified in the protocol that are considered by the investigator to be at least possibly related to therapy with study medications.
Part 1: Maximum Tolerated Dose (MTD) of Orally Administered YK-029A | Cycle 1 (Cycle length is equal to [=] 28 days)
  The MTD is the highest dose level at which the participant tolerates treatment without dose-limiting toxicities.
Part 2: Objective Response Rate (ORR) according to RECIST 1.1 by IRC | Up to 36 months after first dose
  Expansion Cohorts 1、2、3 : Confirmed Objective Response Rate (ORR) Assessed by the Independent Review Committee (IRC)
Part 3: Objective Response Rate (ORR) according to RECIST 1.1 by IRC | Up to 36 months after first dose
  xpansion Cohorts 4、5、6、7、8、9 : Confirmed Objective Response Rate (ORR) Assessed by the Independent Review Committee (IRC)

SECONDARY OUTCOMES:
Part 1:Cmax: Maximum Plasma Concentration for YK-029A and its Active Metabolites after a Single Oral Dose. | Up to 24 hours; Pre-dose and multiple time points post-dose on Cycle 1 Day 1 (C1D1)
Part1:Tmax: Time to Cmax for YK-029A and its Active Metabolites after a Single Oral Dose. | Up to 24 hours; Pre-dose and multiple time points post-dose on C1D1
Part1:AUC24: Area Under the Plasma Concentration-Time Curve from Time 0 to 24 hours for YK-029A and its Active Metabolites after a Single Oral Dose | Up to 24 hours; Pre-dose and multiple time points post-dose on C1D1
Part1:AUClast: Area Under the Plasma Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration for YK-029A and its Active Metabolites after a Single Oral Dose. | Up to 24 hours; Pre-dose and multiple time points post-dose on C1D1
Part1:Cmax, ss: Maximum Plasma Concentration for YK-029A and its Active Metabolites at Steady State after Multiple Oral Doses. | Up to approximately 168 days; Pre-dose and multiple time points post-dose.
Part1:Tmax, ss: Time to Cmax for YK-029A and its Active Metabolites at Steady State after Multiple Oral Doses. | Up to approximately 168 days; Pre-dose and multiple time points post-dose.
AUC24, ss: Area Under the Plasma Concentration-Time Curve from Time 0 to 24 hours for YK-029A and its Active Metabolites at Steady State after Multiple Oral Doses. | Up to approximately 168 days; Pre-dose and multiple time points post-dose.
Part2、3：Overall Response Rate (ORR) as Assessed by the investigator. | Up to 36 months after first dose.
Part2、3：Duration of Response (DOR) | Up to 36 months after first dose.
  Duration of response is defined as the time interval from the time that the measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that PD is objectively documented.
Part2、3：Disease Control Rate (DCR) | Up to 36 months after first dose.
  DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) (in the case of SD, measurements must have met the SD criteria at least once after study entry at a minimum interval of 42 days) after the initiation of study drug.
Part2、3：Progression Free Survival (PFS) | Up to 36 months after first dose.
  PFS is defined as the time interval from the date of randomization until the first date at which the criteria for progressive disease (PD) according to RECIST version 1.1 are met or death, whichever occurs first.
Part2、3：Overall Survival (OS) | Up to 36 months after first dose.
  OS is defined as the interval from the date of randomization until death. OS is defined as the interval from the date of randomization until death. OS is defined as the interval from the date of randomization until death.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhao, Doctor, Study Director — Puhe Biopharma
Locations (35):
- China (35):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanjing, Guangxi
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital Affiliated to Medical School of Nanjing University, Nanjin, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Chest Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - Jilin Tumor Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - the First Affiliated Hospital; Medical College of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Cancer in Zhejiang Province, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Beijing Chest Hospital Affiliated to Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Beijing Tiantan Hospital affiliated to Capital Medical University, Beijing
  - National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - Peking University Cancer Hospital, Beijing
  - The Fifth Medical Center of the Chinese People's Liberation Army General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan J, Wu L, Yang K, Zhao J, Zhao Y, Dai X, Li M, Xie Y, Yao Y, Zhao M, Zhou C, Ren X, Liu Z, Pan Y, Li Y, Liu B, Cheng Y, Miao L, Yu Q, Zhang Z, Liu X, Cui J, Zhang Y, Zhang L, Li X, Li X, Shen B, Chen B, Zeng S, Li B, Hu Y, Li L, Wu R, Song Q, Wang J. Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of YK-029A in Treatment-Naive Patients With Advanced NSCLC Harboring EGFR Exon 20 Insertion Mutations: A Phase 1 Trial. J Thorac Oncol. 2024 Feb;19(2):314-324. doi: 10.1016/j.jtho.2023.09.1449. Epub 2023 Sep 28. PMID 37776953